CLINICAL TRIAL: NCT06382454
Title: Investigation of The Effect of Upper Extremity Robot-Assisted Therapy on Upper Extremity Performance in Stroke Patients
Brief Title: Upper Extremity Robot-Assisted Therapy in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Interact Medical Technologies Inc. (Unknown)
Responsible Party: Principal Investigator, Izel Demirhan, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-5921
Record Dates: First submitted 2024-03-27; First posted 2024-04-24 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Upper Extremity
Keywords: Stroke; Robot-Assisted Therapies; Upper Extremity; Exoskeleton Robot; Motor Performance
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): 30 minutes of individualized trunk, lower extremity and upper extremity exercises; the other 30 minutes will be treated with the robotic system. In the robot-assisted treatment, a total of 12 movements will be used, including the movement patterns that patients have the most difficulty in daily life and two movement patterns used in the Proprioceptive Neuromuscular Facilitation approach. Individual-specific rehabilitation program; individual-specific trunk, lower extremity and upper extremity exercises to be applied in both groups will consist of the following exercises according to the needs of the patients, and the degree of difficulty will be planned according to the needs of the patients. All patients will be treated for 8 weeks, 3 days a week, 60 minutes a day.
  Interventions: Device: Assist-On Arm Robot Group
- Control Group (Active Comparator): For 30 minutes, exercises including trunk, lower extremity and upper extremity exercises specific to the individual will be practiced, while the movement patterns to be used in the robotic system will be practiced in the other 30 minutes with the physiotherapist. Individual-specific rehabilitation program; individual-specific trunk, lower extremity and upper extremity exercises to be applied in both groups will consist of the following exercises according to the needs of the patients, and the degree of difficulty will be planned according to the needs of the patients. All patients will be treated for 8 weeks, 3 days a week, 60 minutes a day.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Assist-On Arm Robot Group — 30 minutes of individualized trunk, lower extremity and upper extremity exercises; the other 30 minutes will be treated with the robotic system. In the robot-assisted treatment, a total of 12 movements will be used, including the movement patterns that patients have the most difficulty in daily life and two movement patterns used in the Proprioceptive Neuromuscular Facilitation approach. Individual-specific rehabilitation program; individual-specific trunk, lower extremity and upper extremity exercises to be applied in both groups will consist of the following exercises according to the needs of the patients, and the degree of difficulty will be planned according to the needs of the patients. All patients will be treated for 8 weeks, 3 days a week, 60 minutes a day.
  Other Names: Assist-On Arm Robot
  Arms: Treatment Group
Other: Control Group — For 30 minutes, exercises including trunk, lower extremity and upper extremity exercises specific to the individual will be practiced, while the movement patterns to be used in the robotic system will be practiced in the other 30 minutes with the physiotherapist. Individual-specific rehabilitation program; individual-specific trunk, lower extremity and upper extremity exercises to be applied in both groups will consist of the following exercises according to the needs of the patients, and the degree of difficulty will be planned according to the needs of the patients. All patients will be treated for 8 weeks, 3 days a week, 60 minutes a day.
  Arms: Control Group

SUMMARY:
Upper extremity hemiparesis is one of the most common symptoms after stroke. Robot-assisted therapies have been used as an approach to rehabilitation of upper extremity hemiplegia in recent years. Robot-assisted therapy is an approach to post-stroke rehabilitation that uses robotic devices to provide motor or task-oriented training to patients. When the literature is examined, there are studies showing that robot-assisted therapies are similar or superior to conventional methods. In order to provide the most effective rehabilitation approach in upper extremity robots, it is suggested that it may be more accurate to consider the robotic device as a training platform consisting of various therapeutic techniques and principles, not as a tool alone. A robotic system will be used to overcome the disadvantages of the existing robotic systems in the literature such as not providing support to the patient at the time of need, not providing fluidity in shoulder movements by not taking into account the scapulohumeral rhythm in upper extremity movements, long installation times, and ignoring task-oriented training. The system to be used is a self-aligning exoskeleton system for robot-assisted upper extremity rehabilitation. The system provides safe and versatile rehabilitation at increasing intensity and also allows for objective assessments. The aim of this clinical study was to evaluate the efficacy of robot-assisted upper limb rehabilitation in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Spasticity of the upper extremity muscles is 2 or less according to the Modified Ashworth Scale
* Stroke patients with a Mini Mental State Examination score of 24 and above will be included in the study

Exclusion Criteria:

* Have a neurological disease other than stroke that may affect upper extremity movements
* Surgery or botox application for upper extremity spasticity in the last 6 months
* History of upper extremity fracture or surgery
* Attending another rehabilitation program
* Individuals who do not agree to participate in the study and do not give written informed consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 5 minutes
  Spasticity of the patients will be evaluated with the Modified Ashworth Scale (MAS). The MAS, which assesses resistance to passive movement, is the most widely used method for the evaluation of muscle tone in the clinic. Spasticity is graded as 0, 1, 1+, 2, 3 and 4 according to the resistance of the muscle.
Fugl-Meyer Assessment Upper Extremity | 15 minutes
  The Fugl Meyer Assessment is a disease-specific assessment designed to evaluate motor function, balance, sensory qualities and joint function in individuals after stroke. The scale consists of 5 sections: motor function, sensory function, balance (standing-sitting), range of motion and joint pain. Scoring is based on the ability to complete each item using a 3-point ordinal scale, where 0 = cannot perform, 1 = partially perform and 2 = fully perform. It is stated in the literature that the scale can also be divided. Therefore, in our study, the upper extremity part of the scale will be used in the evaluation of upper extremity performance before and after treatment. The total score that can be obtained from the Fugl Meyer Upper Extremity assessment is 66 and includes items evaluating joint movements, coordination-speed and reflex activities related to the shoulder, elbow, forearm, wrist and hand.
Action Research Arm Test | 15 minutes
  Action Research Arm Test (ARAT) is a performance-based test that assesses upper extremity skills and functional level. The test has 4 subgroups evaluating coarse grasping, fine grasping, fingertip grasping and gross movement and 19 evaluation items in total. Scoring is between 0 and 3; 0 means 'movement cannot be performed at all' and 3 means 'performance is normal'. For the test, objects of special sizes and shapes suitable for the relevant grasping styles are required.
Box and Block Test | 1 minutes
  The Box and Block Test, which provides a measure of manual dexterity, is administered with two adjacent boxes with a 15.2 cm high partition between them. One of the two boxes, both 53.7 x 25.4 x 8.5 cm in size, is filled with 150 wooden blocks of 2.5 cm3 each. The patient should attempt to move the maximum number of blocks within 60 seconds by grasping each block and carrying it across the compartment to the other compartment.
Nine Hole Peg Test | 10 minutes
  The test consists of a platform with 9 holes and 9 rods. The platform will be placed directly in front of the individuals and the rods will be adjusted so that the rods are on the dominant hand side and the holes are on the non-dominant hand side. After the test rules are explained to the individuals, the individuals will be given the opportunity to practice before the application. Individuals will be asked to insert the rods on the board as fast as possible. The test results will be recorded by measuring the time from the moment the individuals touch the first stick to the moment the last stick is attached to the platform with a stopwatch. Then, they will be asked to remove the 9 bars one by one with the same hand and the removal time will be recorded. The test will be performed for the non-dominant hand using the same method, but this time the platform will be rotated in front of the non-dominant hand.

SECONDARY OUTCOMES:
ACTIVLIM | 5 minutes
  In the scale containing a total of 22 questions, the first 14 questions consist of activities involving adults and children. Questions 15-18 include activities specific to adults and questions 19-22 include activities specific to children. Since the study includes an adult group, the questionnaire including the first 18 questions will be applied to the stroke patients. When applying the ACTIVLIM scale, individuals will be asked to answer by thinking about the last 3 months. This questioning will be done in a way that the individual will be unassisted, independent of the extremity and strategy used. The scale is scored between 0 and 2. "0" means impossible, "1" means difficult, "2" means easy. Activities not performed in the last 3 months are not evaluated and the "question mark (?)" section is marked on the questionnaire page. As a result of the questionnaire, low score means clinically worse activity level and high score means clinically better activity level.
ABILHAND Assessment | 5 minutes
  It is a scale that assesses the manual ability perceived by the individual in daily activities. In our study, the 23-item version of the scale developed for individuals with chronic stroke and including bimanual activities will be used. The scale has 23 items requiring the use of upper extremities and each item is scored as 0: impossible, 1: difficult, 2: easy. Activities not performed in the last 3 months are not scored.
Stroke Impact Scale | 10 minutes
  Stroke Impact Scale 3.0; this scale, which aims to assess the perception of quality of life after stroke by patients themselves or their carers, consists of 8 subsections and 59 questions. Each question is scored by evaluating the difficulty experienced in the last week on a 5-point Likert scale. The score for each section ranges from 0 to 100. In addition to the 8 subsections, it also includes the evaluation of the perception of recovery after stroke with a 0-100 point visual analogue scale (0: No recovery, 100: Full recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Kılınç, Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No